CLINICAL TRIAL: NCT02162030
Title: The Impact of Self as Context in the Treatment of Long-term Health Conditions With Acceptance and Commitment Therapy; a Feasibility Pilot Study
Brief Title: A Component Analysis of Acceptance and Commitment Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Daniel Stockton, Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 139593
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Long-term Physical Health Conditions; Mild to Moderate Anxiety and/or Depression
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full ACT (Other): Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Modified ACT (Other): Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Half of the participants will receive an eight-session ACT intervention whereby each component of the psychological flexibility model will be covered. Half of the participants will receive an eight-session act intervention whereby each component except self as context will be covered.

SUMMARY:
The purpose of this study is to determine whether a specific component of Acceptance and Commitment Therapy (ACT) called 'Self as Context' is an important and necessary part of this therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults of working age (18-65)
* Patients with a primary positive diagnosis of a long-term health condition (The most common conditions referred to the service are Diabetes, Chronic Obstructive Pulmonary Disease [COPD], Rheumatoid Arthritis and Epilepsy) where there is a verifiable medical diagnosis supported by the patients General Practitioner (GP) and/or secondary care physician
* Patients with concurrent mental health difficulties (defined as mild - moderate anxiety and/or depression, see table one).

Exclusion Criteria:

* Patients with a primary diagnosis of 'medically unexplained symptoms' (MUS) including somatoform disorders (e.g. pain disorder, conversion disorder, body dysmorphic disorder, hypochondriasis) and functional somatic syndromes (e.g. irritable bowel syndrome, chronic fatigue syndrome, fibromyalgia, non-cardiac chest pain, non-epileptic seizures)
* Mental health diagnoses in addition to mild - moderate anxiety / depression (e.g. personality disorder, bipolar disorder, psychosis etc.)
* Patients in receipt of secondary care mental health services
* Patients with severe and enduring mental health difficulties
* Significant risk issues, or current substance misuse
* Previous contact with mental health services (defined as two or more prior episodes of contact without significant change)
* Inpatient admission for mental health difficulties within the last five years
* History of overdoses or other self-injury
* Stated reluctance to engage in psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline psychological flexibility at end of 8-session psychological intervention (approximately 8 weeks) and at post-therapy eight week follow-up (using the Acceptance and Action Questionnaire II) | Measure taken at first therapy appointment (baseline), taken again after 8-session intervention (approximately 8 weeks) and again at eight week post-therapy follow-up
  The Acceptance and Action Questionnaire II (Bond et al., 2011) is a 10-item self-report questionnaire measuring psychological flexibility on a 7-point likert scale
Change from baseline self-report 'quality of life' at end of 8-session psychological intervention (approximately 8 weeks) and at post-therapy eight week follow-up (using the Work and Social Adjustment Scale) | Measure taken at first therapy appointment (baseline), taken again after 8-session intervention (approximately 8 weeks) and again at eight week post-therapy follow-up
  The Work and Social Adjustment Scale (Mundt, Marks, Shear, & Greist, 2002) is a 5-item self-report questionnaire measuring functional impairment and disability attributable to the effects of a health condition using a 9-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Stockton, Principal Investigator — University of Sheffield
Locations (1):
- Primary Care Health and Medical Psychology Services, Sheffield, South Yorkshire, United Kingdom